CLINICAL TRIAL: NCT00517166
Title: Survey of Tourniquet Use in a Combat Support Hospital
Status: Completed | Type: Observational
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRAQ 06-010; I.2006.175dt
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Vascular Injury
Keywords: tourniquet; extremity injury; hemostatic device
MeSH Terms: conditions — Vascular System Injuries | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Individuals on whom tourniquet was used.
  Interventions: Device: CAT (Combat Arms Tourniquet)

INTERVENTIONS:
Device: CAT (Combat Arms Tourniquet) — device

SUMMARY:
Data will be collected on the type of tourniquet and circumstances of its use. Patients with penetrating extremity injury will have clinical and pre-clinical hospital data collected.

DETAILED DESCRIPTION:
This is a performance improvement project that is a prospective observational cohort design with subgroup analyses. This project meets the criteria of research with its intent to publish. No data is generated and only existing data are used. No interventions are made and the comparisons will be with within subgroups in the cohort.

Aim 1. Describe the number of tourniquets which were appropriately used (wound required a tourniquet and tourniquet was placed properly) as assessed by treating physician

Aim 2 &3. Describe if limbs wounds with tourniquets were bleeding upon admission, resuscitation, and following tourniquet removal

Aim 4. Describe if mortality for the cohort of patients with tourniquets is different than the mortality predicted by various injury scoring systems

Aim 5. Compare patient outcomes between those in which a tourniquet was indicated but not used and those for whom a tourniquet was indicated and used

Aim 6. Determine if patients that received tourniquets for an extended time period exhibit any known tourniquet complications

ELIGIBILITY:
Inclusion Criteria:

* penetrating extremity injury with tourniquet use

Exclusion Criteria:

* non penetrating extremity injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Combat soldiers on whom tourniquet was applied.
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2006-08; Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Kragh, MD, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- Combat Support Hospital, Baghdad, Iraq

REFERENCES:
- [Derived] Kragh JF Jr, O'Neill ML, Walters TJ, Jones JA, Baer DG, Gershman LK, Wade CE, Holcomb JB. Minor morbidity with emergency tourniquet use to stop bleeding in severe limb trauma: research, history, and reconciling advocates and abolitionists. Mil Med. 2011 Jul;176(7):817-23. doi: 10.7205/milmed-d-10-00417. PMID 22128725
- [Derived] Kragh JF Jr, O'Neill ML, Beebe DF, Fox CJ, Beekley AC, Cain JS, Parsons DL, Mabry RL, Blackbourne LH. Survey of the indications for use of emergency tourniquets. J Spec Oper Med. 2011 Winter;11(1):30-34. doi: 10.55460/36SQ-1UQU. PMID 21455908
- [Derived] Kragh JF Jr, Littrel ML, Jones JA, Walters TJ, Baer DG, Wade CE, Holcomb JB. Battle casualty survival with emergency tourniquet use to stop limb bleeding. J Emerg Med. 2011 Dec;41(6):590-7. doi: 10.1016/j.jemermed.2009.07.022. Epub 2009 Aug 31. PMID 19717268
- [Derived] Kragh JF Jr, Walters TJ, Baer DG, Fox CJ, Wade CE, Salinas J, Holcomb JB. Survival with emergency tourniquet use to stop bleeding in major limb trauma. Ann Surg. 2009 Jan;249(1):1-7. doi: 10.1097/SLA.0b013e31818842ba. PMID 19106667